CLINICAL TRIAL: NCT00150254
Title: A Twelve-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating the Safety and Efficacy of Four Dosing Strategies for CP-526,555 ( 0.5 mg BID Titrated, 0.5 mg BID, 1 mg BID, and Titrated 1 mg BID ) in Smoking Cessation
Brief Title: 12 Week Evaluation of the Safety and Efficacy of 4 Dosing Strategies of CP-526,555 and Placebo for Smoking Cessation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051007
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: CP-526,555 (varenicline)

SUMMARY:
The purpose of the study is to measure the safety and efficacy of four dosing strategies of CP-526,555 for 12 weeks compared with placebo for smoking cessation. Post-treatment follow-up of smoking status to one year from randomization was performed in a non-treatment extension Protocol A3051018

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked on average of at least ten cigarettes per day during the past year
* Subjects must have no period of abstinence greater than three months in the past year

Exclusion Criteria:

* Subjects with any history of clinically significant cardiovascular disease
* Uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625
Dates: Start 2001-09; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
4 week continuous quit rate (CQR) at Weeks 9-12 and Weeks 4-7

SECONDARY OUTCOMES:
Continuous abstinence rate from target quit date to end of treatment (Week 12)
Carbon monoxide(CO)-confirmed 7-day point prevalence of abstinence at Week 12
Number of cigarettes smoked per day
Urge to smoke and withdrawal symptoms assessed by Minnesota Nicotine Withdrawal Scale
Rewarding effects of smoking assessed by Smoking Effects Inventory
Weight change from baselin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Jackson, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051007&StudyName=+12+Week+Evaluation+of+the+Safety+and+Efficacy+of+4+Dosing+Strategies+of+CP%2D526%2C555+and+Placebo+for+Smoking+Cessation%2E